CLINICAL TRIAL: NCT00943176
Title: Modafinil in the Treatment of Fatigue in Patients With Primary Biliary Cirrhosis
Brief Title: Modafinil in the Treatment of Fatigue in Patients With Primary Biliary Cirrhosis (PBC)
Acronym: PBC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Keith D. Lindor, M.D. / PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-007692
Record Dates: First submitted 2009-07-17; First posted 2009-07-22 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Fatigue; Primary Biliary Cirrhosis
Keywords: Fatigue
MeSH Terms: conditions — Fatigue; Liver Cirrhosis, Biliary | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Modafinil
- Modafinil (Experimental)
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — 100 mg tablets of modafinil or matched placebo will be given for a total of 12 weeks. Patients will be instructed to start one capsule once daily (modafinil or placebo), and dose will be titrated according to tolerability and response.
  Other Names: Provigil

SUMMARY:
The purpose of this study is to evaluate the use of modafinil in the treatment of fatigue in patients with Primary Biliary Cirrhosis.

The general aim of the study is to identify a safe and effective therapy for fatigue in patients with primary biliary cirrhosis.

DETAILED DESCRIPTION:
The general aim of the study is to identify a safe and effective therapy for fatigue in patients with primary biliary cirrhosis. Specific aims include: 1) to determine the safety profile of modafinil in patients with primary biliary cirrhosis; 2) to evaluate the beneficial effects of modafinil on patients with primary biliary cirrhosis and fatigue as documented by a well-validated questionnaire (Fisk Fatigue Severity Score) to be applied at the beginning and end of the study period; and 3) to compare the performance of three questionnaires (Fisk Fatigue Severity Score, Fatigue Severity Scale and the fatigue domain of the PBC-40) as instruments to determine the benefits of a therapeutic intervention on fatigue by establishing the minimally important clinical difference of these measures of fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Primary biliary cirrhosis will be defined as present when 2 of 3 of the following criteria are met:

  * Chronic cholestatic liver disease for greater than 6 months with alkaline phosphatase levels greater than 1.5 times the upper limit of normal prior to UDCA treatment.
  * Positive AMA titer greater or equal to 1:40 or AMA greater than 0.1U. Liver histology in the past with features consistent with or diagnostic of PBC.
* A previous ultrasound, computed tomography (CT), or cholangiography of the biliary tree excludes biliary obstruction.
* Verbal report of fatigue for greater than 6 months.

Exclusion Criteria:

* Patients with other serious coexistent conditions such as pre-existing advanced malignancy or severe cardiopulmonary disease which would be expected to limit their expectancy to less than three years.
* Findings highly suggestive of liver disease of other etiology such as chronic alcoholic liver disease, chronic hepatitis B or C infection, hemochromatosis, Wilson's disease, 1-antitrypsin deficiency, non-alcoholic steatohepatitis or sclerosing cholangitis.
* Treatment of underlying PBC has been modified in the preceding six months.
* Anticipated need for transplantation in one year (Mayo survival model <80% one-year survival without transplant) or MELD above 15.
* Recurrent variceal bleeding, presence of diuretic-resistant ascites, or spontaneous encephalopathy.
* Active drug or alcohol use.
* History of drug and/or stimulant (e.g. methylphenidate, amphetamine, or cocaine) abuse.
* Serum bilirubin >4 mg/dl.
* Serum creatinine over 1.4 mg/dl.
* Pregnancy.
* Breast-feeding.
* Inability or unwillingness to practice contraceptive measures for the prevention of pregnancy if appropriate.
* Other fatigue related diagnoses such as anemia, thyroid disease, renal failure, use of beta-blockers and untreated depression.
* Known hypersensitivity to modafinil.
* Uncontrolled hypertension.
* Patients with hypertension and left ventricular hypertrophy documented on ECG in the last 2 years.
* Recent (<6 months) history of myocardial infarction or unstable angina.
* Patients with history of psychosis.
* Patients receiving cyclosporine, warfarin, tricyclic agents, carbamazepine, phenobarbital, rifampin, ketoconazole or itraconazole in the last 3 months.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The main endpoint will be the change in fatigue severity (quantified by the FFSS) following 12 weeks of treatment, compared to baseline values. | after 12 weeks of treatment

SECONDARY OUTCOMES:
Secondary outcome includes frequency of adverse events, change in alkaline phosphatase, AST, total bilirubin and albumin levels after 12 weeks of therapy compared to baseline values, change in fatigue severity compared to baseline. | after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Keith D Lindor, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Silveira MG, Gossard AA, Stahler AC, Jorgensen RA, Petz JL, Ali AH, Lindor KD. A Randomized, Placebo-Controlled Clinical Trial of Efficacy and Safety: Modafinil in the Treatment of Fatigue in Patients With Primary Biliary Cirrhosis. Am J Ther. 2017 Mar/Apr;24(2):e167-e176. doi: 10.1097/MJT.0000000000000387. PMID 27148676